CLINICAL TRIAL: NCT00280072
Title: A Multi-Center, Randomized, Controlled, Double-Blind, Phase II Study To Assess Safety and Efficacy With the Renal Assist Device (RAD) in Patients With Acute Renal Failure
Brief Title: Study to Evaluate the Safety and Efficacy of the Renal Assist Device in Patients With Acute Renal Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: RenaMed Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAD-003
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Kidney Failure, Acute
Keywords: Renal Failure, Acute; Acute Kidney Failure; Acute Renal Failure; Acute Tubular Necrosis; Anuria; Renal Dialysis; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury; Kidney Cortex Necrosis; Anuria

INTERVENTIONS:
Device: Renal Assist Device

SUMMARY:
* The purpose of this study is to evaluate the safety and efficacy of the RAD to determine whether the RAD is effective in reducing mortality in patients with Acute Renal Failure due to Acute Tubule Necrosis and to evaluate the safety of the RAD
* If the RAD works normally when used for as long as 72 hours
* If the RAD will provide added benefits to normal CVVH therapy for patients with Acute Renal Failure

DETAILED DESCRIPTION:
Acute Renal Failure (ARF)is a severe inflammatory disease state often accompanied by Multi-Organ Failure (MOF) and Systemic Inflammatory Response Syndrome (SIRS). ARF is precipitated by many factors and is most often linked to the loss of kidney tubule cell function. Patients with ARF are treated in the intensive care units of hospitals and recovery of renal function is vitally important to their survival. Current therapy for ARF involves conventional kidney support with continuous renal replacement therapies (CRRT). Despite advances in treating patients with CRRT, ARF has an extremely high mortality rate (55-70%) and requires extensive hospital stays, predominantly in the ICU. The RAD is designed to both treat ARF with MOF and/or SIRs and facilitate the natural recovery of a patient's own kidney function. The RAD is intended for use for short periods of time in conventional extracorporeal therapeutic systems that are already available in the hospital. The RAD therapy operates outside the body, and is designed to mimic the structure and function of the natural kidney. In this manner it is intended to replace the missing metabolic, endocrine, and immunologic functions of the kidney and allow time for the patient's own kidneys to resume normal functions.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Acute Tubular Necrosis (ATN)
* At least one non-renal organ failure

Exclusion Criteria:

* A renal transplant at any time
* Chronic renal failure occurring due to reasons other than Acute Tubular Necrosis (ATN)
* Chronic
* Chronic immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate all cause mortality at Day 28

SECONDARY OUTCOMES:
To assess the effect of RAD treatment in measures of patient's safety and clinical outcome

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - Denver Nephrologists, PC, Denver, Colorado
  - George Washington University Hospital, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - WNERTA, Springfield, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Southeast Renal Associates, Charlotte, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Texas, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia